CLINICAL TRIAL: NCT04647591
Title: ENT Barotrauma Epidemiology Among French Army Divers
Brief Title: Diver Ear, Nose and Throat Barotrauma Epidemiology
Acronym: BTORL PAF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Direction Centrale du Service de Santé des Armées (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2020PRI07; 2020-A02893-36 (Other: Id-RCB)
Record Dates: First submitted 2020-10-23; First posted 2020-12-01 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Barotrauma Epidemiology
Keywords: ENT barotrauma; Epidemiology; Risk factors; Diving; Professional impact; Barotrauma management
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ENT Barotrauma incidence and link with risk factors (Experimental)
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — Use of a questionnaire focused on diver experience and medical history upon inclusion and another questionnaire in case of ENT Barautrauma over a period of two years to standardize Barotrauma assessment.

SUMMARY:
Ear, nose and throat barotrauma are the most frequently encountered accidents during diving. One study related to recreational diving reports that ENT barotrauma concern 10% of dives with experimented divers and 30% with novice divers. Nevertheless, a low number of studies were realized on ENT barotrauma, particularly those involving middle ear and sinuses, maybe because most of them evolve favorably without sequelae.

Besides, it has been described that pathologies which may induce chronic or acute tubal dyspermeability can result in an increased middle ear or sinus barotrauma risk. But once again no study was realized which objective was to look for an association between these risk factors and for the association strength between risk factors and ENT barotrauma occurrence. Few data on military population exist either. However, operational constraints, stressing environment with necessity of realizing performances to validate diving certificate or other military diving specificities can lead one to think that military divers have an increased risk to be subjected to ENT barotrauma. Furthermore, therapeutic measures and more particularly physicians' attitude concerning a temporary incapacity period to avoid recurrence or clinical worsening of barotrauma differ depending on diving centers. But the question to resume diving or not is essential for military staff given that temporary incapacity may lead to training cessation or can be questioned because of operational constraints requiring anticipated diving resumption.

The purpose of this research is to study middle ear and sinus barotrauma thanks to questionnaires focused on those pathologies and their potential risk factors. The hypothesis is that it will allow identification of main risk factors in order to develop preventive measures as well as the characteristics and missions of concerned divers and the impact of those barotrauma on this population.

DETAILED DESCRIPTION:
Ear, nose and throat barotrauma are the most frequently encountered accidents during diving. It has been described that pathologies which may induce chronic or acute tubal dyspermeability can result in an increased middle ear or sinus barotrauma risk. But no study was realized which objective was to look for an association between these risk factors and for the association strength between risk factors and ENT barotrauma occurrence.

Futhermore, few data on military population exist while operational constraints, stressing environment with necessity of realizing performances to validate diving certificate or other military diving specificities can lead one to think that military divers have an increased risk to be subjected to ENT barotrauma. Therapeutic measures and more particularly physicians' attitude concerning a temporary incapacity period to avoid recurrence or clinical worsening of barotrauma differ depending on diving centers. But the question to resume diving or not is essential for military staff given that temporary incapacity may lead to training cessation or can be questioned because of operational constraints requiring anticipated diving resumption.

The aim of this research is then to study middle ear and sinus barotrauma in order to identify main risk factors, the characteristics and missions of concerned military divers and the impact of those pathologies on this population. Two kind of questionnaires will be used : one which will be completed by divers just after their inclusion in the study and one that will be filled in case of ENT barotrauma suspicion over a period of two years. The first questionnaire will give information about diving level and medical history and the second one will allow standardized assessment of barotrauma suspicion . Divers will be followed for two years, whether they experience an ENT barotrauma or not.

ELIGIBILITY:
Inclusion Criteria:

* French military professional diver of French army diver following diving training (this includes navy, land forces, police, air force, army health service)
* 18 year or older man or woman

Exclusion Criteria:

* Diver opposing his study participation
* Diver who doesn't master enough French language reading or understanding to be able to oppose his study participation
* Every other reason which, according to investigator, might interfere with the assessment of research outcomes
* Diver being part of special forces

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-10-04 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
ENT Barotrauma incidence among French army divers and student divers followed for 2 years | 4 years
  Number of ENT barotrauma occurring among French army divers and student divers enrolled in the study for 2 years. Characteristics of concerned divers (diving level, medical history…) will also be presented. ENT Barotrauma events will be defined according to Haines and Harris classification after otoscopic examination for middle ear and by sinus pain sudden onset during diving for sinuses. Clinical confirmation will be obtained through questioning and suggestive disease history. In case of doubt, a scanner will be used.

SECONDARY OUTCOMES:
Correlation between ENT barotrauma and divers characteristics | 4 years
  Correlation will be performed between ENT events and characteristics of enrolled divers (diving level, dive kind, medical history…) to determine if one these characteristics constitutes a risk factor
ENT barotrauma treatment | 4 years
  Treatments prescribed for ENT barotrauma will be presented.
ENT barotrauma-induced incapacity periods | 4 years
  Duration of incapacity periods that will be prescribed after ENT barotrauma events will be presented.
ENT barotrauma incidence among student divers followed for one year | 3 years
  Number of ENT barotrauma occurring among French army student divers enrolled in the study and followed for 1 year. Characteristics of concerned student divers (diving level, medical history…) will also be presented. ENT Barotrauma events will be defined according to Haines and Harris classification after otoscopic examination for middle ear and by sinus pain sudden onset during diving for sinuses. Clinical confirmation will be obtained through questioning and suggestive disease history. In case of doubt, a scanner will be used.
ENT barotrauma-induced permanent incapacities | 4 years
  Number of permanent incapacities induced by ENT barotrauma will be presented.

CONTACTS AND LOCATIONS:
Overall Officials: Jean Morin, MD, Study Director — Hopital d'Instruction des Armées Sainte Anne
Locations (7):
- France (7):
  - 160e Antenne Médicale d'Antibes, Antibes, Alpes Maritimes
  - 2nd Groupe Plongeurs Démineurs Brest, Brest, Finistère
  - 1er Groupe Plongeurs Démineurs Cherbourg, Cherbourg, Manche
  - 152e Antenne Médicale de St Mandrier, Toulon, Var
  - 3e Groupe Plongeurs Démineurs Toulon, Toulon, Var
  - Base navale de Toulon, Toulon, Var
  - Service de médecine hyperbare et expertise de la plongée, Toulon, Var

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Taylor DM, O'Toole KS, Ryan CM. Experienced scuba divers in Australia and the United States suffer considerable injury and morbidity. Wilderness Environ Med. 2003 Summer;14(2):83-8. doi: 10.1580/1080-6032(2003)014[0083:esdiaa]2.0.co;2. PMID 12825881
- [Background] Fitzpatrick DT, Franck BA, Mason KT, Shannon SG. Risk factors for symptomatic otic and sinus barotrauma in a multiplace hyperbaric chamber. Undersea Hyperb Med. 1999 Winter;26(4):243-7. PMID 10642071
- See also: Related Info — https://www.editions-ellipses.fr/accueil/2064-physiologie-et-medecine-de-la-plongee-9782729829834.html